CLINICAL TRIAL: NCT02304770
Title: A Pilot Study of Aminolaevulinic Acid (ALA) Photodynamic Therapy (PDT) in Patients With Cervical Persistent High Risk HPV Infection or Cervical Intraepithelial Neoplasia
Brief Title: Aminolaevulinic Acid Photodynamic Therapy of Cervical Persistent HPV Infection and Cervical Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDZJALA-201409
Record Dates: First submitted 2014-11-23; First posted 2014-12-02 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Cervical Persistent High Risk HPV Infection; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- cervical persistent high risk HPV infection (Experimental): Aminolaevulinic acid photodynamic therapy for the treatment of patients with cervical persistent high risk HPV infection
  Interventions: Drug: Aminolaevulinic acid photodynamic therapy
- CIN 1 with high risk HPV infection (Experimental): Aminolaevulinic acid photodynamic therapy for the treatment of patients with CIN 1 and high risk HPV infection
  Interventions: Drug: Aminolaevulinic acid photodynamic therapy
- CIN 2/3 (Experimental): Aminolaevulinic acid photodynamic therapy for the treatment of patients with CIN 2/3
  Interventions: Drug: Aminolaevulinic acid photodynamic therapy

INTERVENTIONS:
Drug: Aminolaevulinic acid photodynamic therapy — Aminolaevulinic acid mediated photodynamic therapy

SUMMARY:
The study will examine the effect of aminolaevulinic acid (ALA) photodynamic therapy (PDT) of cervical precancerous lesions in women.

ELIGIBILITY:
Inclusion Criteria:

1. Premenopausal women, 25-50 years of age
2. Meet one of the 3 following conditions:

   high-risk HPV-DNA persistently positive for at least 6 months, without CIN or higher grade lesions as verified by cervical biopsy within the last 3 months; CIN1 as verified by cervical biopsy within the last 3 months and high-risk HPV-DNA positive; CIN2/3 as verified by cervical biopsy within the last 3 months, with intense desire to retain the cervical structure or function
3. Satisfactory colposcopy examination (visibility of entire transformation zone and entire lesion margin ) and endocervical curettage negative
4. In good health condition as confirmed by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis on the screening and baseline evaluation within the last 4 weeks of the onset of the study
5. Meet the following conditions: pregnancy test negative; no pregnancy plan during the trial;no sexuality or reliable contraceptive measures taken since last menstruation to the onset of the study, agreeing to adopt reliable contraceptive measures during the study
6. Written informed consent signed

Exclusion Criteria:

1. Atypical glandular cells of undetermined significance (AGUS) or adenocarcinoma in situ (AIS) on cytology ,or malignant cells on cytology or histology, or other suspicion of either micro-invasive or invasive disease
2. Invasive carcinoma possibility or positive endocervical curettage on colposcopy
3. Severe pelvic inflammatory disease, severe cervicitis, or other severe gynaecological infection as per clinical examination
4. Undiagnosed vaginal bleeding
5. With allergic disease at present; known or suspected porphyria; known allergy to ALA or similar compounds
6. Evidence or history of clinically significant cardiovascular, endocrine, neurologic, pulmonary, hematological, immunological, psychiatric, metabolic disease or other serious diseases
7. Pregnancy or nursing
8. Therapeutic drug or other therapeutic measures applied on cervix or rectum within the last 2 weeks of the onset of the study
9. Participation in any clinical studies within the last 30 days
10. Subjects that the investigators judged to be not suitable to participate the study besides above

Ages: 25 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Response Rate | 3 months after treatments
  Based on histology
clearance of high risk HPV | 3 months after treatments
  proportion of patients with high risk HPV clearance

CONTACTS AND LOCATIONS:
Overall Officials: Beihua Kong, MD, Principal Investigator — Qilu Hospital of Shandong University; Youzhong Zhang, MD, Principal Investigator — Qilu Hospital of Shandong University; Jining Tao, Master, Study Director — Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd.
Locations (4):
- China (4):
  - The First Affliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang